CLINICAL TRIAL: NCT01835080
Title: Effect of Pulmonary Arterial Hypertension Treatment on Obstructive Sleep Apnea
Brief Title: Obstructive Sleep Apnea (OSA) in Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Inova Health Care Services (Other)
Collaborators: Brown University (Other); Tufts University (Other); George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: 12.038
Record Dates: First submitted 2013-04-10; First posted 2013-04-18 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2014-06

CONDITIONS: Pulmonary Arterial Hypertension; Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea, ,; Pulmonary Arterial Hypertension; sleep study,; polysomnogram,; Respiratory Disturbance Index (RDI)
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether pulmonary arterial hypertension can worsen or even cause sleep apnea. It is hypothesized that if pulmonary arterial hypertension does indeed worsen or cause sleep apnea, then the treatment should first focus on the underlying pulmonary arterial hypertension instead of the sleep apnea.

To determine if a person has sleep apnea, they will undergo one overnight polysomnogram (sleep study). If it is found that they have mild to moderate sleep apnea, then the subject will be invited to continue in the study and their pulmonary arterial hypertension will be treated by their managing primary physician. After the subject has had treatment for their pulmonary arterial hypertension, the study center will have them return for a follow up sleep study to learn the effects of pulmonary arterial hypertension treatment management on their sleep apnea, 12-24 weeks after the first sleep study.

DETAILED DESCRIPTION:
Pulmonary Arterial Hypertension (PAH) is associated with fluid retention. Currently, the treatment paradigm for newly diagnosed PAH patients includes evaluation for Obstructive Sleep Apnea (OSA). The investigators propose that untreated or sub-optimally managed PAH patients have significant fluid retention which redistributes to the upper body during sleep and exacerbates or even mimics OSA. The investigators hypothesize that treatment of PAH patients with vasodilators and diuretics to optimize fluid balance will attenuate or even resolve OSA prior to the initiation of specific therapy for OSA (CPAP).

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of Group 1 PAH

  * Either lack of treatment for PAH or sub-optimally treated PAH as defined by NYHA FC 3 or 4
  * Age 18 or older
  * Ability to give consent
  * Ability to undergo overnight polysomnogram
  * Previously diagnosed OSA not on therapy

Exclusion Criteria:

* Age younger than 18
* Pregnancy
* Previously diagnosed OSA and receiving therapy
* Inability to undergo overnight polysomnography in laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosis of Group 1 PAH Either lack of treatment for PAH or sub-optimally treated PAH
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is a decrease in Respiratory Disturbance Index (RDI) by 10 events/hour | 12-24 weeks
  All patients will undergo a sleep study (polysomnogram) before their PAH is treated (or treated optimally) and each patient will have a repeat sleep study at 12- 24 weeks after their PAH treatment is optimally managed by their primary managing physician. These sleep studies will be centrally scored to determine whether a decrease in RDI of at least 10 events/hour has been met.

SECONDARY OUTCOMES:
Decrease in neck circumference by 0.9 cm | 12-24 weeks
  All subjects will be assessed for decrease in neck circumference by 0.9 cm
Decrease in ankle circumference by 0.8 cm | 12-24 weeks
  All subjects will be assessed for decrease in ankle circumference by 0.8 cm
improvement in Epworth Sleepiness Scale | 12-24 weeks
  All subjects will be assessed for improvement in Epworth Sleepiness Scale
improvement in Arousal Index | 12-24 weeks
  All subjects will be assessed for improvement in Arousal Index

CONTACTS AND LOCATIONS:
Overall Officials: Nargues Weir, MD, Principal Investigator — NIH/Inova Fairfax Hospital
Locations (1):
- Inova Heart and Vascular Institute/Inova Fairfax Hospital, Falls Church, Virginia, United States

REFERENCES:
- [Background] Proceedings of the 4th World Symposium on Pulmonary Hypertension, February 2008, Dana Point, California, USA. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S1-117. No abstract available. PMID 19630151
- [Background] Bady E, Achkar A, Pascal S, Orvoen-Frija E, Laaban JP. Pulmonary arterial hypertension in patients with sleep apnoea syndrome. Thorax. 2000 Nov;55(11):934-9. doi: 10.1136/thorax.55.11.934. PMID 11050263
- [Background] Ulrich S, Fischler M, Speich R, Bloch KE. Sleep-related breathing disorders in patients with pulmonary hypertension. Chest. 2008 Jun;133(6):1375-1380. doi: 10.1378/chest.07-3035. Epub 2008 Mar 13. PMID 18339776
- [Background] Badesch DB, Raskob GE, Elliott CG, Krichman AM, Farber HW, Frost AE, Barst RJ, Benza RL, Liou TG, Turner M, Giles S, Feldkircher K, Miller DP, McGoon MD. Pulmonary arterial hypertension: baseline characteristics from the REVEAL Registry. Chest. 2010 Feb;137(2):376-87. doi: 10.1378/chest.09-1140. Epub 2009 Oct 16. PMID 19837821
- [Background] Brown LM, Chen H, Halpern S, Taichman D, McGoon MD, Farber HW, Frost AE, Liou TG, Turner M, Feldkircher K, Miller DP, Elliott CG. Delay in recognition of pulmonary arterial hypertension: factors identified from the REVEAL Registry. Chest. 2011 Jul;140(1):19-26. doi: 10.1378/chest.10-1166. Epub 2011 Mar 10. PMID 21393391
- [Background] Atwood CW Jr, McCrory D, Garcia JG, Abman SH, Ahearn GS; American College of Chest Physicians. Pulmonary artery hypertension and sleep-disordered breathing: ACCP evidence-based clinical practice guidelines. Chest. 2004 Jul;126(1 Suppl):72S-77S. doi: 10.1378/chest.126.1_suppl.72S. PMID 15249496
- [Background] Redolfi S, Arnulf I, Pottier M, Lajou J, Koskas I, Bradley TD, Similowski T. Attenuation of obstructive sleep apnea by compression stockings in subjects with venous insufficiency. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1062-6. doi: 10.1164/rccm.201102-0350OC. PMID 21836140
- [Background] Friedman O, Bradley TD, Chan CT, Parkes R, Logan AG. Relationship between overnight rostral fluid shift and obstructive sleep apnea in drug-resistant hypertension. Hypertension. 2010 Dec;56(6):1077-82. doi: 10.1161/HYPERTENSIONAHA.110.154427. Epub 2010 Nov 8. PMID 21060007
- [Background] Elias RM, Bradley TD, Kasai T, Motwani SS, Chan CT. Rostral overnight fluid shift in end-stage renal disease: relationship with obstructive sleep apnea. Nephrol Dial Transplant. 2012 Apr;27(4):1569-73. doi: 10.1093/ndt/gfr605. Epub 2011 Nov 5. PMID 22058175
- [Background] Redolfi S, Arnulf I, Pottier M, Bradley TD, Similowski T. Effects of venous compression of the legs on overnight rostral fluid shift and obstructive sleep apnea. Respir Physiol Neurobiol. 2011 Mar 15;175(3):390-3. doi: 10.1016/j.resp.2011.01.001. Epub 2011 Jan 8. PMID 21220055
- [Background] Jafari B, Mohsenin V. Overnight rostral fluid shift in obstructive sleep apnea: does it affect the severity of sleep-disordered breathing? Chest. 2011 Oct;140(4):991-997. doi: 10.1378/chest.11-0044. Epub 2011 Mar 24. PMID 21436243